CLINICAL TRIAL: NCT03224767
Title: Phase II Trial of BRAF/MEK Inhibitors in Papillary Craniopharyngiomas
Brief Title: Vemurafenib and Cobimetinib in Treating Patients With BRAF V600E Mutation Positive Craniopharyngioma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A071601; NCI-2017-00740 (Registry Identifier: NCI Clinical Trial Reporting Program); U10CA180821 (NIH)
Record Dates: First submitted 2017-07-19; First posted 2017-07-21 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-01

CONDITIONS: BRAF V600E Mutation Present; Papillary Craniopharyngioma
MeSH Terms: conditions — Craniopharyngioma | interventions — Vemurafenib; cobimetinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (vemurafenib, cobimetinib) (Experimental): Patients receive vemurafenib PO BID on day 1-28 and cobimetinib PO QD on days 1-21. Treatment repeats every 28 days for up to 5 courses in the absence of disease progression or unacceptable toxicity. Patients may then receive radiation therapy, surgery, or continued treatment with vemurafenib and cobimetinib at the discretion of the treating physician.
  Interventions: Drug: Vemurafenib; Drug: Cobimetinib; Other: Laboratory Biomarker Analysis; Other: Quality-of-Life Assessment

INTERVENTIONS:
Drug: Vemurafenib — Given PO
Drug: Cobimetinib — Given PO
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Quality-of-Life Assessment — Ancillary studies

SUMMARY:
This phase II trial studies how well vemurafenib and cobimetinib work in treating patients with BRAF V600E mutation positive craniopharyngioma. Vemurafenib and cobimetinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the activity of BRAF and MEK inhibitor combination in untreated papillary craniopharyngiomas as measured by best response at any time during the first four cycles of BRAF and MEK inhibitor treatment.

II. To determine the activity of BRAF and MEK inhibitor combination in papillary craniopharyngiomas that have progressed after prior radiation treatment with or without surgical resection as measured by best response at any time during the first four cycles of BRAF and MEK inhibitor treatment.

SECONDARY OBJECTIVES:

I. To determine the progression-free survival of patients with papillary craniopharyngiomas receiving BRAF and MEK inhibitors.

II. To determine the toxicity of BRAF/MEK inhibitors in patients with papillary craniopharyngiomas.

III. To determine the activity of BRAF and MEK inhibitor combination in papillary craniopharyngiomas as measured by response of enhancing volume of craniopharyngioma.

IV. To determine the activity of BRAF and MEK inhibitor combination in papillary craniopharyngiomas as measured by response of nonenhancing volume of craniopharyngioma.

V. To determine the overall survival of patients with papillary craniopharyngiomas receiving BRAF and MEK inhibitors.

VI. To determine the duration of response in patients with papillary craniopharyngiomas receiving BRAF and MEK inhibitors.

TERTIARY OBJECTIVES:

I. To evaluate visual fields in patients with papillary craniopharyngiomas who have received BRAF/MEK inhibitors.

II. To evaluate pituitary hormone replacement over time in patients with papillary craniopharyngiomas who have received BRAF/MEK inhibitors.

III. To evaluate the time to response in patients with papillary craniopharyngiomas receiving BRAF and MEK inhibitors.

IV. To assess toxicity that may be associated with radiotherapy in patients with papillary craniopharyngiomas who have received BRAF/MEK inhibitors.

V. To evaluate molecular biomarkers of response in papillary craniopharyngiomas.

VI. To evaluate circulating tumor cells and cell-free circulating deoxyribonucleic acid (DNA) in patients with papillary craniopharyngiomas.

OUTLINE:

Patients receive vemurafenib orally (PO) twice daily (BID) on day 1-28 and cobimetinib PO once daily (QD) on days 1-21. Treatment repeats every 28 days for up to 5 courses in the absence of disease progression or unacceptable toxicity. Patients may then receive radiation therapy, surgery, or continued treatment with vemurafenib and cobimetinib at the discretion of the treating physician.

After completion of study treatment, patients with disease progression are followed up every 16 weeks for 2 years and all other patients are followed up every 6 months for 5 years.

ELIGIBILITY:
* Pre-registration: Patients must have local diagnosis of papillary craniopharyngioma and have tissue slides available for submission to central pathology review; central pathology review will include immunohistochemistry (IHC) testing for BRAF V600E mutation (VE1 clone) and beta-catenin IHC (membranous, non-nuclear pattern) if needed to confirm diagnosis of papillary craniopharyngioma
* Histologically proven papillary craniopharyngioma as documented by central pathology review with positive BRAF V600E mutation by IHC
* Measurable disease and/or non-measurable disease

  * Measurable disease, defined as bidimensionally measurable lesions with clearly defined margins by magnetic resonance imaging (MRI) scans, with a minimum diameter of 10 mm in both dimensions
  * Progressive disease required in cohort B, defined as an increase in the bidirectional area by 25% within the past 13 months after surgery or radiation; progressive or recurrent disease is not required in cohort A, but is allowed provided it is a new diagnosis and patient has not received prior treatment.
* Prior treatment

  * Cohort A: No prior therapy received other than surgery
  * Cohort B: Prior radiation therapy required (any type of prior radiation is allowed)

    * For patients treated with external beam radiation therapy, interstitial brachytherapy or radiosurgery, an interval of >= 3 months must have elapsed from completion of radiation therapy to registration
    * Recovered to Common Terminology Criteria for Adverse Events (CTCAE) grade 1 or less toxicity attributed to radiation with exception of alopecia, fatigue
  * For patients enrolling on Cohort A or Cohort B:

    * For patients treated with surgery, an interval of >= 21 days must have elapsed prior to registration
    * No prior treatment with BRAF or MEK inhibitors
    * Steroid dosing stable for at least 4 days prior to registration
* Not pregnant and not nursing; for women of childbearing potential only, a negative pregnancy test done =< 7 days prior to registration is required
* ECOG performance status =< 2
* Comorbid conditions

  * No evidence of active bleeding, bleeding diathesis, or hemoptysis (>= 1/2 teaspoon of red blood) =< 8 weeks prior to registration
  * No evidence of intracranial hemorrhage =< 4 weeks prior to registration
  * Patients who have experienced thromboembolic event within 6 months prior to registration must be on stable therapeutic anticoagulation for at least 4 weeks prior to registration
  * No symptomatic congestive heart failure (New York Heart Association class II, III, or IV) within 6 months prior to registration
  * No current unstable angina or uncontrolled arrhythmia
  * No uncontrolled hypertension at time of registration (blood pressure [BP] > 150/95 despite antihypertensive therapy)
  * No known history of prolonged QT syndrome
  * No known history of ventricular arrhythmia within 6 months of registration
  * No known history of uveitis or iritis =< 4 weeks prior to registration
  * No known history of or evidence of retinal pathology that is considered a risk factor for neurosensory retinal detachment, retinal vein occlusion (RVO), or neovascular macular degeneration within 12 months of registration
  * No known history of chronic lung disease
* Concomitant medications

  * Chronic concomitant treatment with strong CYP3A4 inducers or CYP3A4 inhibitors is not allowed; patients must discontinue the drug at least 14 days prior to study registration
  * Chronic concomitant treatment with CYP1A2 substrate is not allowed; patients must discontinue the drug at least 14 days prior to study registration
* Absolute neutrophil count >= 1500/mm^3
* Platelets >= 100,000/mm^3
* Creatinine =< 1.5 mg/dL OR creatinine clearance >= 45mL/min
* Bilirubin =< 1.5 upper limit of normal (ULN)
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) =< 2.5 ULN

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-01-05 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
Response rate | Up to 5 years
  Defined as the number of responses achieved during treatment with BRAF and MEK inhibitors divided by the total number of evaluable patients and assessed by contrast-enhanced magnetic resonance imaging or computed tomography. Point estimates will be generated for response rates within each cohort with corresponding 95% binomial confidence intervals. Simon's two-stage design with one interim analysis for futility will be applied to evaluate response rate within each cohort.

SECONDARY OUTCOMES:
Progression-free survival | Up to 5 years
  Will be summarized for each cohort within each cohort with Kaplan-Meier curves and estimates.
Overall survival | Up to 5 years
  Will be summarized for each cohort within each cohort with Kaplan-Meier curves and estimates.

CONTACTS AND LOCATIONS:
Overall Officials: Priscilla K. Brastianos, MD, Study Chair — Massachusetts General Hospital
Locations (106):
- United States (106):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Sutter Cancer Centers Radiation Oncology Services-Auburn, Auburn, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Mills-Peninsula Medical Center, Burlingame, California
  - Sutter Cancer Centers Radiation Oncology Services-Cameron Park, Cameron Park, California
  - Eden Hospital Medical Center, Castro Valley, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Memorial Medical Center, Modesto, California
  - Palo Alto Medical Foundation-Camino Division, Mountain View, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - Sutter Cancer Centers Radiation Oncology Services-Roseville, Roseville, California
  - Sutter Roseville Medical Center, Roseville, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Palo Alto Medical Foundation-Sunnyvale, Sunnyvale, California
  - Sutter Cancer Centers Radiation Oncology Services-Vacaville, Vacaville, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - Smilow Cancer Center/Yale-New Haven Hospital, New Haven, Connecticut
  - Yale University, New Haven, Connecticut
  - Smilow Cancer Hospital Care Center-Trumbull, Trumbull, Connecticut
  - Mayo Clinic in Florida, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Tampa General Hospital, Tampa, Florida
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Idaho Urologic Institute-Meridian, Meridian, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Rush University Medical Center, Chicago, Illinois
  - Central Care Cancer Center - Garden City, Garden City, Kansas
  - Central Care Cancer Center - Great Bend, Great Bend, Kansas
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Corewell Health Grand Rapids Hospitals - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Trinity Health Muskegon Hospital, Muskegon, Michigan
  - Corewell Health Lakeland Hospitals - Niles Hospital, Niles, Michigan
  - Cancer and Hematology Centers of Western Michigan - Norton Shores, Norton Shores, Michigan
  - Corewell Health Reed City Hospital, Reed City, Michigan
  - Corewell Health Lakeland Hospitals - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Corewell Health Lakeland Hospitals - Saint Joseph Hospital, Saint Joseph, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Minnesota Oncology - Burnsville, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Fairview Clinics and Surgery Center Maple Grove, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - Monticello Cancer Center, Monticello, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Rutgers New Jersey Medical School, Newark, New Jersey
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Cancer Centers of Southwest Oklahoma Research, Lawton, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - M D Anderson Cancer Center, Houston, Texas
  - Farmington Health Center, Farmington, Utah
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - South Jordan Health Center, South Jordan, Utah
  - Inova Schar Cancer Institute, Fairfax, Virginia
  - FHCC South Lake Union, Seattle, Washington
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - University of Washington Medical Center - Montlake, Seattle, Washington
  - United Hospital Center, Bridgeport, West Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Camden Clark Medical Center, Parkersburg, West Virginia
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Welch Cancer Center, Sheridan, Wyoming

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Brastianos PK, Twohy E, Geyer S, Gerstner ER, Kaufmann TJ, Tabrizi S, Kabat B, Thierauf J, Ruff MW, Bota DA, Reardon DA, Cohen AL, De La Fuente MI, Lesser GJ, Campian J, Agarwalla PK, Kumthekar P, Mann B, Vora S, Knopp M, Iafrate AJ, Curry WT Jr, Cahill DP, Shih HA, Brown PD, Santagata S, Barker FG 2nd, Galanis E. BRAF-MEK Inhibition in Newly Diagnosed Papillary Craniopharyngiomas. N Engl J Med. 2023 Jul 13;389(2):118-126. doi: 10.1056/NEJMoa2213329. PMID 37437144
- [Derived] Rutenberg MS, Rotondo RL, Rao D, Holtzman AL, Indelicato DJ, Huh S, Morris CG, Mendenhall WM. Clinical outcomes following proton therapy for adult craniopharyngioma: a single-institution cohort study. J Neurooncol. 2020 Apr;147(2):387-395. doi: 10.1007/s11060-020-03432-9. Epub 2020 Feb 21. PMID 32086697